CLINICAL TRIAL: NCT06600373
Title: Study on the Intervention of Mindfulness-integrated Volleyball Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ye Zhiyin (Other)
Responsible Party: Sponsor-Investigator, Ye Zhiyin, Teaching assistant, Central University of Finance and Economics, China
Organization: Central University of Finance and Economics, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUFinanceEcon
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-10

CONDITIONS: Depression, Anxiety; Mindful Walking Meditation
Keywords: mindfulness walking; volleyball; sport therapy
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Conduct approximately 10 minutes of mindful walking after the 110-minute regular physical education group class.
  Interventions: Behavioral: Mindful Walking meditation
- Control group (Active Comparator): 120 minutes regular physical education group class.
  Interventions: Behavioral: physical education group class

INTERVENTIONS:
Behavioral: Mindful Walking meditation — Conduct approximately 10 minutes of mindful walking after the 110-minute regular physical education group class.
  Arms: Experimental group
Behavioral: physical education group class — 120 minutes physical education group class about volleyball.
  Arms: Control group

SUMMARY:
The purpose of this clinical trial is to understand whether a mindfulness-integrated volleyball team sports program can effectively intervene in the mental health of college students, and whether it has better intervention effects compared to a regular volleyball team sports program. The main questions it aims to answer are:

Does the mindfulness-integrated volleyball team sports program effectively intervene in the participants' mental health levels, including indicators such as anxiety and depression? The researchers will compare the mindfulness-integrated volleyball team sports program with the regular volleyball team sports program to see if the intervention effects are more effective.

Participants will:

Attend a mindfulness-integrated volleyball team sports program once a week for 2 hours each session, for a total of 16 weeks.

Complete a psychological questionnaire at the beginning and the end of the program concludes.

DETAILED DESCRIPTION:
The study will focus on a non-clinical population of college students, using an exploratory parallel randomized controlled trial design. Based on the inclusion criteria, participants will be allocated to the experimental group and control group according to their registration time. The experimental group will receive the mindfulness-integrated volleyball program, while the control group will participate in a regular volleyball program. The intervention will last for a total of 16 weeks, with sessions held once a week for 120 minutes each. Relevant assessments will be conducted at two time points: on the day before the intervention, and on the last day of the intervention.

Primary indicators: Youth version of the Patient Health Questionnaire, Generalized Anxiety Disorder Scale.

Secondary indicators: Insomnia Severity Index, Self-Efficacy Scale, Positive and Negative Affect Scale, Life Satisfaction Scale, Self-Esteem Scale, Self-Compassion Scale, Loneliness Scale, Social Anxiety Scale, Perceived Social Support Scale.

All of the above indicators will be measured using the corresponding questionnaires at two time points: T1 pre-test (before the start), T2 after 16 weeks of intervention, for a total of two assessments.

Inclusion criteria: (1) Participants aged ≥16 years; (2) Able to communicate in Mandarin and willing to voluntarily participate in this study; (3) Agree to consistently attend each mindfulness-integrated volleyball session.

Exclusion criteria: (1) Individuals with language communication barriers or unwilling to cooperate in this study; (2) Individuals unable to commit to attending each mindfulness-integrated volleyball session.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 16 years or older.
* Able to communicate in Mandarin and voluntarily participate in the study.
* Agree to consistently participate in each mindfulness-integrated volleyball course.

Exclusion Criteria:

* Disagree to consistently participate in each mindfulness-integrated volleyball course.
* Individuals unable to commit to participating in each mindfulness-integrated volleyball course.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-03-02 (Actual); Study Completion 2025-03-02 (Actual)

PRIMARY OUTCOMES:
depression | From enrollment to the end of treatment at 16 weeks
  Using GAD-7 to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2(after 16 weeks of intervention).
anxiety | From enrollment to the end of treatment at 16 weeks
  Using PHQ-9 to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2 (after 16 weeks of intervention).
social anxiety | From enrollment to the end of treatment at 16 weeks
  Using Mini-SPIN to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2(after 16 weeks of intervention).
insomnia | From enrollment to the end of treatment at 16 weeks
  Using ISI-7 to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2(after 16 weeks of intervention).
positive and negative affects | From enrollment to the end of treatment at 16 weeks
  Using PANAS to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2(after 16 weeks of intervention).
life satisfaction | From enrollment to the end of treatment at 16 weeks
  Using SWLS to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2(after 16 weeks of intervention).

SECONDARY OUTCOMES:
self-esteem | From enrollment to the end of treatment at 16 weeks
  Using WFI to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2(after 16 weeks of intervention).
self-efficacy | From enrollment to the end of treatment at 16 weeks
  Using GSES to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2(after 16 weeks of intervention).
self compassion | From enrollment to the end of treatment at 16 weeks
  Using SCS-SF to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2(after 16 weeks of intervention).
loneliness | From enrollment to the end of treatment at 16 weeks
  Using Revised ULS-3 to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2(after 16 weeks of intervention).
perceived support | From enrollment to the end of treatment at 16 weeks
  Using BPSSQ to investigate the psychological variables of participants, a total of two assessments will be conducted, including T1 pre-test (before the start) and T2(after 16 weeks of intervention).

CONTACTS AND LOCATIONS:
Locations (1):
- Central University of Finance and Economics, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided